CLINICAL TRIAL: NCT03566446
Title: A Phase-1-first in Man Study in Patients With CALR-mutant Myeloproliferative Neoplasms by Vaccinating With CALR Exon 9 Mutant Peptide
Brief Title: CALR Exon 9 Mutant Peptide Vaccine to Patients With CALR-mutant Myeloproliferative Neoplasms
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, Professor, MD, PhD, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPN1801; 2018-000132-10 (EudraCT Number)
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Myeloproliferative Neoplasm, Unclassifiable; Essential Thrombocythemia; Myelofibrosis
Keywords: CALR mutation
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 36 aminoacid CALR exon 9 mutated peptide (Experimental): 15 vaccines, over the course of 1 year
  Interventions: Biological: CALRLong36 peptide

INTERVENTIONS:
Biological: CALRLong36 peptide — 200 ug CALRLong36 peptide in water mixed with 500ul montanide

SUMMARY:
A phase-I-first in man study in patients with calreticulin(CALR)-mutant MPN by vaccinating with exon 9 mutated peptide with the adjuvant Montanide ISA-51 to monitor safety and toxicity and the immunological response to vaccination.

DETAILED DESCRIPTION:
The Philadelphia-chromosome negative chronic myeloproliferative neoplasms (MPN) are acquired cancer diseases, that arise due to mutations in the hematopoietic stem cells in the bone marrow. Median age at diagnosis is approximately 65 years of age and approximately 400 Danes are diagnosed with MPN annually. The MPN comprise essential thrombocythemia (ET), polycythemia vera (PV) and primary myelofibrosis (PMF). In December 2013 two independent research groups reported on the occurrence of somatic mutations in exon 9 of the calreticulin gene in patients with ET and PMF.

The overall rationale for a vaccine with CALR-mutant epitopes is that it will initiate a CALR-mutant specific immune response, which will "release the brakes" on the CALR-mutant specific immune response.

10 patients treated with standard therapy are needed for the trial and each patient will receive 15 vaccinations over the course of one year.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of essential thrombocythemia, post essential thrombocythemia myelofibrosis, prefibrotic myelofibrosis or primary myelofibrosis according to the World Health Organization criteria33 2. Verified mutation in CALR exon 9. 4. Performance status ≤ 2 (ECOG-scale) 5. Expected survival > 3 months 6. Sufficient bone marrow function, i.e.

1. Leucocytes ≥ 1,5 x 109
2. Granulocytes ≥ 1,0 x 109
3. Thrombocytes ≥ 20 x 109
4. Hemoglobin ≥ 7 mmol/L 7. Creatinine < 2.5 upper normal limit, i.e. < 300 µmol/l 8. Sufficient liver function, i.e.

a. Alanine aminotransferase < 2.5 upper normal limit, i.e. ALAT <112 U/l b. Bilirubin < 30 U/l 9. For women: Agreement to use contraceptive methods with a failure rate of < 1% per year during the treatment period and for at least 120 days after the last treatment.

10. For men: Agreement to use contraceptive measures and agreement to refrain from donating sperm.

Exclusion Criteria:

1. Other malignancies in the medical history excluding squamous cell carcinoma. Patients cured for another malignant disease with no sign of relapse three years after ended treatment is allowed to enter the protocol.
2. Significant medical condition per investigators judgement e.g. severe Asthma/chronic obstructive pulmonary disease , poorly regulated heart condition, insulin dependent diabetes mellitus.
3. Acute or chronic viral or bacterial infection e.g. HIV, hepatitis or tuberculosis
4. Serious known allergies or earlier anaphylactic reactions.
5. Known sensibility to Montanide ISA-51
6. Any active autoimmune diseases e.g. autoimmune neutropenia, thrombocytopenia or hemolytic anemia, systemic lupus erythematosus, scleroderma, myasthenia gravis, autoimmune glomerulonephritis, autoimmune adrenal deficiency, autoimmune thyroiditis etc.
7. Pregnant and breastfeeding women.
8. Fertile women not using secure contraception with a failure rate less than < 1%
9. Patients taking immune suppressive medications incl. corticosteroids and methotrexate at the time of enrollment
10. Psychiatric disorders that per investigator judgment could influence compliance.
11. Treatment with other experimental drugs
12. Treatment with other anti-cancer drugs - except interferon (IFN)-a, hydroxyurea or anagrelide.
13. Treatment with ruxolitinib.
14. Treatment with chemotherapy or immune therapy (excluding IFN-a, hydroxyurea or anagrelide) within the last 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Adverse events evaluated by CTCAE 4.03 | 1 year
  Adverse events are graded 1-5 according to the criteria

SECONDARY OUTCOMES:
Immune responses | 1 year
  T-cell cytokine release towards target antigens

OTHER OUTCOMES:
Mutational status | 1 year
  CALR-mutational status
Bone marrow response | 1 year
  bone marrow description
mutational landscape change | 1 year
  Next Generation Sequencing pre- and post-treatment
Overall response | 1 year
  Revised response criteria by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) and European LeukemiaNet (ELN) consensus report

CONTACTS AND LOCATIONS:
Overall Officials: Jacob H Grauslund, MD, Principal Investigator — Center for Cancer Immune Therapy, Denmark
Locations (1):
- Herlev Hospital, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handlos Grauslund J, Holmstrom MO, Jorgensen NG, Klausen U, Weis-Banke SE, El Fassi D, Schollkopf C, Clausen MB, Gjerdrum LMR, Breinholt MF, Kjeldsen JW, Hansen M, Koschmieder S, Chatain N, Novotny GW, Petersen J, Kjaer L, Skov V, Met O, Svane IM, Hasselbalch HC, Andersen MH. Therapeutic Cancer Vaccination With a Peptide Derived From the Calreticulin Exon 9 Mutations Induces Strong Cellular Immune Responses in Patients With CALR-Mutant Chronic Myeloproliferative Neoplasms. Front Oncol. 2021 Feb 26;11:637420. doi: 10.3389/fonc.2021.637420. eCollection 2021. PMID 33718228